CLINICAL TRIAL: NCT00454792
Title: Rehabilitation of Patients With Modic Changes in the Lumbar Spine - a Randomized Controlled Trial
Brief Title: Rehabilitation of Patients With Modic Changes in the Lumbar Spine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Back Research Center, Denmark (Other)
Collaborators: Velux Fonden (Other)
Responsible Party: Principal Investigator, Rikke Krüger Jensen, MSc, The Back Research Center, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VF-20060111
Record Dates: First submitted 2007-03-30; First posted 2007-04-02 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Low Back Pain
Keywords: Low back pain; Modic changes
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise and advise to stay active (Active Comparator): The exercise group received exercises for the stabilising muscles in the low back and abdomen together with dynamic exercises, exercises for postural instability and light physical fitness training.
  Interventions: Other: Exercise
- Rest and use of flexible lumbar belt (Experimental): The rest group was instructed to avoid hard physical activity and to rest twice daily for one hour, by lying down
  Interventions: Other: Restitution

INTERVENTIONS:
Other: Exercise — Back exercise: At home every day. In groups once a week. Duration 10 weeks.
  Arms: Exercise and advise to stay active
Other: Restitution — Restitution: At home 2 times one hour. Meetings every 2 weeks. Duration 10 weeks.
  Arms: Rest and use of flexible lumbar belt

SUMMARY:
The purpose of this study is to compare patients with low back pain (LBP) and Modic Changes from The Backcenter Funen, Ringe:

1. To compare the effect of two types of non-operative treatments:

   A. exercise and advice to be physically active

   B. restitution and advice not to overload the spine
2. To investigate if the results of the treatment are influenced by gender, age, smoking, and physical load.

DETAILED DESCRIPTION:
The clinical experience is that many patients with Modic changes have relatively severe and persistent LBP, which typically appears to be resistant to treatment. Furthermore, a retrospective study at The Backcenter Funen, Ringe, shows that patients with MC fail to improve engaging physical activity. This is unfortunate, because the typical rehabilitation for patients with persistent LBP is back exercises and information about keeping physically active. This means that this relatively large subgroup of patients with Modic changes probably does not improve with the rehabilitation tools used today.

A randomised controlled trial has therefore been designed to study the specific subgroup of patients with Modic changes. In this study we will compare the present "state-of-the art" rehabilitation approach to persistent LBP (namely to exercise and keep active) with a new concept (restitution). The justification for this is that restitution reduces mechanical stress on the vertebrae and therefore would allow heeling of the possible micro fractures in Modic changes.

ELIGIBILITY:
Inclusion Criteria:

Primary inclusion criteria for receiving MRI

* The patient must have LBP with a current duration of 3 - 12 month.
* The patient must have an actual pain intensity ≥4 on numerical pain rating scale from 0-10.

Secondary inclusion criteria for receiving MRI

* The patient must speak and understand Danish.
* The patient must be between 18-60 years of age.
* The patient must be willing to participate in the project. Inclusions criterium for the project
* There must be an MRI showing MC in the lumbar spine.

Exclusion Criteria:

* The patient is unable to go through with the project because of other physical or mental disorder.
* The patient is pregnant.
* The patient is referred to operation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2007-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is actual LBP, as measured with an "11 point box scale". | 10 weeks and 12 months

SECONDARY OUTCOMES:
General Health, as measured with the EQ-5D (EuroQol) | 10 weeks and 12 months
General improvement, as measured with two global instruments a 7-point transition question and an assessment score consisting of a "bothersomeness index" | 10 weeks and 12 months
Physical functions measured with "Roland Morris Disability Questionnaire" | 10 weeks and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Claus Manniche, Prof.Dr.Med., Study Chair — Spine Centre of Southern Denmark
Locations (1):
- Spine Centre of Southern Denmark, Middelfart, Denmark

REFERENCES:
- [Derived] Jensen RK, Leboeuf-Yde C, Wedderkopp N, Sorensen JS, Manniche C. Rest versus exercise as treatment for patients with low back pain and Modic changes. A randomized controlled clinical trial. BMC Med. 2012 Feb 29;10:22. doi: 10.1186/1741-7015-10-22. PMID 22376791